CLINICAL TRIAL: NCT05784948
Title: Efficacy of Virtual Reality Mindfulness in Patients With Psychosis
Brief Title: Safety and Efficacy of Virtual Reality Mindfulness in Patients With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-01-042
Record Dates: First submitted 2023-02-08; First posted 2023-03-27 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia Spectrum Disorders; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Psychotic Disorder Not Otherwise Specified
Keywords: Virtual Reality Mindfulness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Mindfulness Treatment (Experimental): Experience virtual reality mindfulness treatment with a screen from a head-mounted display for 30 minutes in a comfortable sitting position.
  Interventions: Other: Virtual Reality Mindfulness Treatment
- Relaxing scenery and music experience (Sham Comparator): Experience relaxing scenery and music with a screen from a head-mounted display for 30 minutes in a comfortable sitting position.
  Interventions: Other: Experience relaxing scenery and music

INTERVENTIONS:
Other: Virtual Reality Mindfulness Treatment — once a week for 30 minutes, over 8 weeks
  Arms: Virtual Reality Mindfulness Treatment
Other: Experience relaxing scenery and music — once a week for 30 minutes, over 8 weeks
  Arms: Relaxing scenery and music experience

SUMMARY:
This study is to evaluate the safety and efficacy of Virtual Reality Mindfulness in Patients With Psychosis.

DETAILED DESCRIPTION:
This study is randomized, single-blind and parallel group trial to evaluate the safety and the efficacy of Virtual Reality Mindfulness in Patients With Psychosis once a week over 8 weeks treatment period. Both groups can experience the screen coming out of the head-mounted display for 30 minutes in a comfortable sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 15-59 years (inclusive) of age at time of consent.
* Patients with current DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-fifth edition) diagnosis schizophrenia spectrum and other psychotic disorders including bipolar and related disorders or depressive disorder with psychotic symptoms.
* Patients who can agree to participate in the study in a stable state (Clinical Global Impression score of 5 or less) and cooperate appropriately with questionnaires and tests.
* Patients with a SOFAS score in the range of 41 to 80 points.
* Patients with a PANSS score of less than 85 points.

Exclusion Criteria:

* Patients who are currently in poor health due to serious physical illness
* Patients who are currently pregnant or lactating.
* Patients who are accompanying intellectual disability with an Intelligence Quotient (IQ) of 70 or lower
* Patients who have difficulty in agreeing to and participating in research due to severely impaired ability to verify reality
* Patients with a PANSS score of 85 or higher or a CGI of 6 or higher
* Patients with a SOFAS score of 40 or less or 81 or more
* Patients who are currently in hospitalized

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessment by Experience Questionnaire Decentering | 1 week
  The experience questionnaire (EQ) is a psychological measure used to assess attentional bias.
  The questionnaire consists of 15 items, with a minimum score of 1 and a maximum score of 7. The higher scores indicate the better outcome.

SECONDARY OUTCOMES:
Efficacy Assessment by Psychotic Symptom Rating Scales (PSYRATS) | 1 week
  Korean Psychotic Symptom Rating Scales-Delision (K-PSYRATS-D) is to assess whether the assessed individual is experiencing delusional symptoms. This subscale consists of 11 items, with a minimum score of 0 (none) and a maximum score of 4 (extremely severe). The total score for this subscale ranges from 0 to 44, with a minimum score of 0 and a maximum score of 44. The higher scores indicate more severe delusional symptoms.
Efficacy Assessment by Psychotic Symptom Rating Scales (PSYRATS) | 1 week
  Korean Psychotic Symptom Rating Scales-Auditory Hallucination (K-PSYRATS-AH) is used to assess the presence of hallucination symptoms in the individual being evaluated. This subscale consists of 11 items, with a minimum score of 0 (none) and a maximum score of 4 (extremely severe). Higher scores indicate more severe hallucination symptoms.
Efficacy Assessment by Korea-Polyenvironmental Risk Score-I (PERS-I) | through study completion, an average of 8 weeks
  Korea-PERS-I assesses the risk of developing psychosis based on six factors: paternal age at birth, parental socioeconomic status (SES), urbanicity, childhood trauma, adult life events, and clinical high-risk state for psychosis. Paternal age over 35 years is scored as 0.5 if exposed and -0.5 if not. Parental SES is scored as 1 if receiving medical aid and 0 if not. Urbanicity is scored as 0 for living in a city and -3 for not. Childhood trauma is scored as 4.5 if exposed and 0 if not. Adult life events are scored as 5.5 if exposed and -2 if not. Clinical high-risk state for psychosis is scored as 10 if exposed and 0 if not. The scores for all six factors are added up to obtain a total score, with higher scores indicating greater risk. Data will be collected twice, one week before and after the intervention.
Efficacy Assessment by Korea-Polyenvironmental Risk Score-II (PERS-II) | through study completion, an average of 8 weeks
  Korea-PERS-II assesses the risk of developing psychosis based on six factors: paternal age at birth, obstetric complications, parental SES, urbanicity, childhood adversity, and recent life events. Paternal age is scored based on age ranges, with scores ranging from 0 to 2. Obstetric complications are scored as 2 if birth weight is less than 2.5kg and 0 if not. Parental SES is scored based on income and education levels, with scores ranging from -1.5 to 3. Urbanicity is scored based on living location, with scores ranging from -2 to 0.5. Childhood adversity includes neglect, emotional abuse, physical abuse, and sexual abuse, with scores ranging from 0 to 5.5. Sexual abuse with moderate levels is scored as 4 if exposed and 0 if not. Recent life events are scored as 3 if exposed and -2 if not. The scores for all six factors are added up to obtain a total score, with higher scores indicating greater risk. Data will be collected twice, one week before and after the intervention.
Efficacy Assessment by Positive and Negative Syndrome Scale | 1 week
  Positive and Negative Syndrome Scale (PANSS) is a scale used to assess the severity of positive, negative, and cognitive symptoms in patients with psychotic disorders, minimum of each item (Positive Scale, Negative Scale and General Psychopathology Scale) is 1, maximum is 7. The higher number is worse outcome. The data will be taken twice, i.e., within one-week before and after the intervention.
Efficacy Assessment by Social and Occupational Functioning Assessment Scale | 1 week
  Social and Occupational Functioning Assessment Scale (SOFAS) consists of ranging from 100 points (excellent functioning) to 0 points (grossly impaired functioning). The specific rating criteria for SOFAS are as follows: Self-care, Social functioning, Occupational functioning, Educational functioning, Leisure functioning. The higher scores indicating higher levels of functioning. The data will be taken twice within one-week before and after the intervention.
Efficacy Assessment by Health of the Nation Outcome Scales | 1 week
  Health of the Nation Outcome Scales (HoNOS) is a scale used to assess the mental health and social functioning of patients. It consists of 12 items, minimum of each item is 0, maximum is 4. The higher scores indicate more severe patient conditions. The data will be taken twice within one-week before and after the intervention.
Efficacy Assessment by Columbia-Suicide Severity Rating Scale | 1 week
  Columbia-Suicide Severity Rating Scale (C-SSRS) is a scale used to assess suicide risk. It includes 9 items, minimum of each item is 0, maximum is 4. The higher scores indicating greater risk. The data will be taken twice within one-week before and after the intervention.
Safety Assessment by Skin conductance level | 1 week
  Skin conductance level (SCL) results are typically expressed in microsiemens (μS), which is the unit of electrical conductivity. The range of skin conductance level values is usually 0.5~50 μS, under conditions of emotional excitement, anxiety, and tension, leading to an increase in skin conductance level.
Safety Assessment by Heart rate | 1 week
  Heart rate (HR) is the number of times the heart beats per minute and is typically measured in beats per minute (bpm). The resting heart rate for adults is generally between 60-100 bpm. A higher heart rate typically indicates that the heart needs to beat faster to meet the body's needs, which may be caused by factors such as emotional excitement, exercise, stress, pain, or illness.
Safety Assessment by R-R interval | 1 week
  The R-R interval is the time interval between adjacent R waves on an electrocardiogram (ECG) and is typically measured in seconds. The normal range of the R-R interval is usually between 0.6-1.2 seconds. A higher RR interval typically indicates an abnormal heart rhythm or some form of heart problem.
Efficacy Assessment by self rating scale Perceived Stress Scale (PSS) | 1 week
  The Perceived Stress Scale (PSS) consists of 10 items, with each item rated on a 5-point scale ranging from 0 (never) to 4 (very often). The minimum score on the scale is 0, and the maximum score is 40. The higher scores on the PSS indicate higher levels of perceived stress. The data will be taken twice within one-week before and after the intervention.
Efficacy Assessment by self rating scale Subjective Wellbeing under Neuroleptics(SWN-K) | 1 week
  Subjective Wellbeing under Neuroleptics (SWN-K) consists of 20 questions. The minimum score for each question is zero and the maximum score is five. The reverse scoring questions include 1,4,6,9,10,11,12,14,16,17. The total score of the whole item is obtained, and the lower the score, the worse the subjective well-being. The data will be taken twice within one-week before and after the intervention.
Efficacy Assessment by self rating scale Motivation and Pleasure Scale-Self Report (MPS-SR) | 1 week
  The Motivation and Pleasure Scale-Self Report (MPS-SR) consists of 14 questions, each rated on a 10-point scale, where the minimum and maximum scores for each item are 0 and 10, respectively, with higher scores indicating greater levels of motivation and pleasure. The data will be taken twice within one-week before and after the intervention.
Efficacy Assessment by self rating scale Beck Depression Inventory (BDI) | 1 week
  Beck Depression Inventory (BDI) consists of 21 items including cognitive, emotional, synchronous, and physical symptoms of depression. The total score ranges from 0~63 points for each question. Its score is 0 ~ 9 points non-depression, 10 ~ 15 is mild depression, 16 ~ 23 is moderate depression, and 24 ~ 63 is severe depression. The data will be taken twice within one-week before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Department of Psychiatry, Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea